CLINICAL TRIAL: NCT01687166
Title: Clinical Evaluation of the Blazer Open-Irrigated Ablation Catheter for the Treatment of Paroxysmal Atrial Fibrillation
Acronym: ZERO-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDM00048665
Record Dates: First submitted 2012-08-29; First posted 2012-09-18 (Estimated); Results first posted 2018-06-18 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Paroxysmal Atrial Fibrillation (PAF)
Keywords: Paroxysmal Atrial Fibrillation; Cardiac Arrhythmias; Heart Disease; Cardiovascular Disease; Radiofrequency Ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blazer Open-Irrigated Ablation Catheter (Experimental): Blazer Open-Irrigated Ablation Catheter and Ablation Catheter Cable used in conjunction with a compatible electroanatomic mapping system
  Interventions: Device: Blazer Open-Irrigated Ablation Catheter (Boston Scientific)
- FDA Approved Open-Irrigated Ablation Catheter (Active Comparator): FDA approved Open-Irrigated Radiofrequency Ablation Catheter system and compatible electroanatomic mapping system for the treatment of paroxysmal atrial fibrillation.
  Interventions: Device: FDA Approved Open-Irrigated Ablation Catheter

INTERVENTIONS:
Device: Blazer Open-Irrigated Ablation Catheter (Boston Scientific)
  Arms: Blazer Open-Irrigated Ablation Catheter
Device: FDA Approved Open-Irrigated Ablation Catheter
  Arms: FDA Approved Open-Irrigated Ablation Catheter

SUMMARY:
The purpose of this study is to establish the safety and effectiveness of the Blazer Open-Irrigated radiofrequency ablation catheter for the treatment of drug refractory, recurrent, symptomatic, paroxysmal atrial fibrillation.

DETAILED DESCRIPTION:
The ZERO-AF trial is a prospective, multicenter, single blind, 1:1 randomized study. The trial is designed to demonstrate that the safety and effectiveness of the Blazer® Open-Irrigated Ablation Catheter are non-inferior to the safety and effectiveness of the control catheters, for the treatment drug refractory, recurrent, symptomatic, paroxysmal atrial fibrillation. The control catheters are open-irrigated radiofrequency ablation catheters that are approved in the United States for the treatment of drug refractory recurrent symptomatic paroxysmal atrial fibrillation, when used with compatible three-dimensional electroanatomic mapping systems.

ELIGIBILITY:
Inclusion Criteria:

* History of recurrent symptomatic PAF with ≥2 episodes reported within the 365 days prior to enrollment

  o PAF is AF episodes that last ≥30 seconds in duration and terminate within 7 days.
* At least 1 episode of PAF documented by Holter monitor, rhythm strip, trans-telephonic monitor (TTM), or 12-lead ECG in the 365 days prior to enrollment
* Refractory to at least one Beta Blocker, Calcium Channel Blocker, Class I OR Class III anti-arrhythmic drug (AAD)
* Age 18 or above, or of legal age to give informed consent specific to state and national law
* Competent and willing to provide written informed consent to participate in the study and agree to comply with follow-up visits and evaluation

Exclusion Criteria:

* Have any of the following heart conditions within 90 days prior to enrollment:

  * New York Heart Association (NYHA) Class III or IV
  * Left ventricular ejection fraction (LVEF) <35%
  * Left atrial (LA) diameter >5.5 cm
  * Unstable angina or ongoing myocardial ischemia
  * Transmural myocardial infarction (MI)
* Congenital structural heart disease that increases the risk of ablation or precludes catheter placement
* Undergone any left atrial catheter or surgical ablation
* Have had a coronary intervention, cardiac surgery, or other cardiac ablation within 90 days prior to enrollment
* Had >1 AF episode lasting greater than 7 days, with no episodes having lasted greater than 30 days, within the past year
* Subjects regularly prescribed amiodarone therapy during the 120 days prior to enrollment
* Contraindication to anticoagulation therapy
* Creatinine >2.5mg/dl or creatinine clearance <30mL/min within 90 days (3 months) prior to enrollment
* Prosthetic mitral or tricuspid heart valves
* Confirmed cardiac thrombus within 30 days (1 month) prior to enrollment
* Implanted pacemaker, ICD, or CRT leads within 180 days (6 months) prior to enrollment
* History of CVA, TIA or PE within 180 days (6 months) prior to enrollment
* Left atrial appendage closure device
* Any other significant uncontrolled or unstable medical condition (e.g. sepsis, acute metabolic illness, end stage COPD)
* Enrolled in any concurrent clinical trial without documented pre-approval from BSC
* Women who are pregnant or plan to become pregnant within the course of their participation in the investigation
* Life expectancy ≤ 2 years (730 days) per physician opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Actual)
Dates: Start 2012-10; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Natale, M.D., Principal Investigator — Texas Cardiac Arrhythmia Institute at St. David's Medical Center
Locations (38):
- United States (27):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Hunstville Hospital, Huntsville, Alabama
  - Sequoia Hospital, Redwood City, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - St. Vincent's Medical Center, Jacksonville, Florida
  - Baptist Hospital, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Georgia Health Sciences University, Augusta, Georgia
  - Union Memorial Hospital, Baltimore, Maryland
  - Caritas St. Elizabeth's Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - New York University, New York, New York
  - Mt. Sinai Medical Center, New York, New York
  - Strong Memorial Hospital of the University of Rochester, Rochester, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Trinity Mother of Frances Health System, Tyler, Texas
  - University of Virginia, Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
- Australia (2):
  - Heart Care Partners, Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Na Homolce Hospital, Prague, Czechia
- CHU of Bordeaux, Pessac, Gironde, France
- Germany (2):
  - Charité University Berlin, Berlin
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
- Centro Hospital de Santa Cruz, Carnaxide, Portugal
- Spain (2):
  - Hospital Clinico Y Provincial, Barcelona
  - Clínica Universitaria de Navarra, Pamplona
- Karolinska University Hospital, Stockholm, Sweden
- Golden Jubilee National Hospital, Glasgow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Blazer Open-Irrigated Ablation Catheter: Blazer Open-Irrigated Ablation Catheter and Ablation Catheter Cable used in conjunction with a compatible electroanatomic mapping system
  Blazer Open-Irrigated Ablation Catheter (Boston Scientific)
- Control: FDA approved Open-Irrigated Radiofrequency Ablation Catheter system and compatible electroanatomic mapping system for the treatment of paroxysmal atrial fibrillation.
  FDA Approved Open-Irrigated Ablation Catheter
- Blazer Open-Irrigated Ablation Catheter Roll-In: Blazer Open-Irrigated Ablation Catheter Roll-In Subjects (Not randomized)
- Control Roll-In: Non-Randomized Subjects treated with an FDA approved Open-Irrigated Radiofrequency Ablation Catheter system and compatible electroanatomic mapping system for the treatment of paroxysmal atrial fibrillation.
  FDA Approved Open-Irrigated Ablation Catheter
Period: Overall Study
Arm/Group | Blazer Open-Irrigated Ablation Catheter | Control | Blazer Open-Irrigated Ablation Catheter Roll-In | Control Roll-In
Started | 167 | 172 | 56 | 3
Completed | 139 | 145 | 42 | 1
Not Completed | 28 | 27 | 14 | 2
Not completed — Attempt subject | 2 | 3 | 2 | 0
Not completed — Did not meet eligibility criteria | 4 | 6 | 1 | 1
Not completed — Adverse Event | 2 | 1 | 0 | 0
Not completed — Physician Decision | 3 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 4 | 3 | 0
Not completed — Lost to Follow-up | 2 | 5 | 1 | 0
Not completed — Equipment/Device Availability | 0 | 1 | 0 | 0
Not completed — Death | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 0
Not completed — Subject moved out of state | 0 | 1 | 0 | 0
Not completed — Patient unable to be compliant | 1 | 0 | 0 | 0
Not completed — Physician choice to use different device | 1 | 2 | 4 | 0
Not completed — Insurance | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blazer Open-Irrigated Ablation Catheter | Control | Blazer Open-Irrigated Ablation Catheter Roll-In | Control Roll-In | Total
Number analyzed (Participants) | 167 | 172 | 56 | 3 | 398
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11) | 59 (10) | 62 (10) | 61 (10) | 60 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 65 | 15 | 1 | 143
  Male | 105 | 107 | 41 | 2 | 255
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 0 | 1 | 0 | 0 | 1
  United States | 107 | 112 | 46 | 2 | 267
  United Kingdom | 3 | 3 | 1 | 0 | 7
  Australia | 6 | 5 | 2 | 0 | 13
  France | 3 | 3 | 0 | 0 | 6
  Portugal | 3 | 2 | 3 | 1 | 9
  Germany | 18 | 18 | 0 | 0 | 36
  Spain | 27 | 28 | 4 | 0 | 59
Height [Mean (Standard Deviation); unit: cm] | 173 (9) | 174 (9) | 175 (11) | 175 (11) | 174 (10)
Weight [Mean (Standard Deviation); unit: kg] | 89 (19) | 90 (22) | 94 (21) | 79 (15) | 90 (21)
Resting Heart Rate [Mean (Standard Deviation); unit: bpm] | 71 (19) | 67 (15) | 68 (17) | 68 (7) | 69 (17)
New York Heart Assessment (NYHA) Class [Count of Participants; unit: Participants] — NYHA Class at enrollment based upon the following definitions:
  Class I - Subjects with heart disease who are able to remain at a comfortable state while performing ordinary physical activity Class II - Subjects who are comfortable at rest or with mild exertion but experience symptoms with more strenuous activity Class III - Subjects who are comfortable at rest but experience symptoms with mild activity Class IV - Subjects who are symptomatic at rest and are unable to carry out any physical activity
  Participants
    I | 67 | 64 | 20 | 3 | 154
    II | 17 | 13 | 10 | 0 | 40
    Non Heart Failure (HF) | 76 | 92 | 24 | 0 | 192
    Not Assessed | 7 | 3 | 2 | 0 | 12

OUTCOME MEASURES:

1. Primary Outcome: Procedure-related Complication Free Rate
Description: The safety of the Blazer OI catheter will be evaluated by demonstrating that the investigational group serious adverse event rate is non-inferior to that of the control group.
  The safety of the Blazer OI catheter will be evaluated by demonstrating that the investigational group rate of significant pulmonary vein stenosis (≥70% reduction in diameter from baseline) and atrio-esophageal fistulas is non-inferior to that of the control group.
Time Frame: 12 Months
Population: Outcome Measures were not assessed for the non-randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Blazer Open-Irrigated Ablation Catheter | Control
Number analyzed (Participants) | 157 | 164
Participants | 140 | 148

2. Primary Outcome: Chronic Success Rate
Description: The primary effectiveness of the Blazer OI catheter will be evaluated by demonstrating that the proportion of subjects free from failure* in the investigational group is non-inferior to those in the control group.
  *failure is defined as a randomized subject being an acute procedural failure, having more than one repeat procedure during the 90 day blanking period or having a documented symptomatic atrial fibrillation, atrial tachycardia, atrial fibrillation between 91 days and 12 months post-procedure.
Time Frame: Within 12 months of the index procedure
Population: Outcome Measures were not assessed for the non-randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Blazer Open-Irrigated Ablation Catheter | Control
Number analyzed (Participants) | 157 | 164
Participants | 102 | 108

3. Secondary Outcome: Acute Success
Description: Demonstration that the investigational group acute procedural success rate is non-inferior to that of the control group. Acute procedural success is defined as a subject that successfully had all clinically relevant veins electrically isolated, by demonstration of entrance block at a minimum and no evidence of exit conduction with the randomized investigational or control catheter only.
Time Frame: Acute- During Index Procedure, 20 minutes after confirmation of Pulmonary Vein Isolation
Population: Outcome Measures were not assessed for the non-randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Blazer Open-Irrigated Ablation Catheter | Control
Number analyzed (Participants) | 157 | 164
Participants | 155 | 163

ADVERSE EVENTS:
Time Frame: Adverse events were collected from enrollment to end of follow-up ~12Months.
Description: Adverse event data is reported for treatment and attempt subjects.
Groups:
- Blazer Open-Irrigated Ablation Catheter Randomized: Blazer Open-Irrigated Ablation Catheter and Ablation Catheter Cable used in conjunction with a compatible electroanatomic mapping system
  Blazer Open-Irrigated Ablation Catheter (Boston Scientific)
- FDA Approved Open-Irrigated Ablation Catheter Randomized: FDA approved Open-Irrigated Radiofrequency Ablation Catheter system and compatible electroanatomic mapping system for the treatment of paroxysmal atrial fibrillation.
  FDA Approved Open-Irrigated Ablation Catheter
- Blazer Open-Irrigated Ablation Catheter Roll-In: Roll-In Cases for Blazer Open-Irrigated Ablation Catheter and Ablation Catheter Cable used in conjunction with a compatible electroanatomic mapping system
  Blazer Open-Irrigated Ablation Catheter (Boston Scientific)
- FDA Approved Open-Irrigated Ablation Catheter Roll-In: Roll-In Cases for FDA approved Open-Irrigated Radiofrequency Ablation Catheter system and compatible electroanatomic mapping system for the treatment of paroxysmal atrial fibrillation.
  FDA Approved Open-Irrigated Ablation Catheter
Arm/Group | Blazer Open-Irrigated Ablation Catheter Randomized | FDA Approved Open-Irrigated Ablation Catheter Randomized | Blazer Open-Irrigated Ablation Catheter Roll-In | FDA Approved Open-Irrigated Ablation Catheter Roll-In
All-Cause Mortality (participants affected / at risk) | 1/159 | 1/167 | 0/51 | 0/1
Serious Adverse Events (participants affected / at risk) | 66/159 | 65/167 | 19/51 | 0/1
Other Adverse Events (participants affected / at risk) | 104/159 | 95/167 | 33/51 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blazer Open-Irrigated Ablation Catheter Randomized (N=159) | FDA Approved Open-Irrigated Ablation Catheter Randomized (N=167) | Blazer Open-Irrigated Ablation Catheter Roll-In (N=51) | FDA Approved Open-Irrigated Ablation Catheter Roll-In (N=1)
AV Fistula (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Adverse medication reaction (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alcohol dependency (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Ablation Procedure) (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Atrial fibrillation (AF) (Cardiac disorders) | 18 (18) | 27 (28) | 6 (6) | 0 (0)
Atrial flutter (type 1 Isthmus Dependent) (Cardiac disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Atypical Atrial Flutter (Cardiac disorders) | 5 (6) | 2 (2) | 1 (1) | 0 (0)
Atypical atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cancer (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade/perforation (Cardiac disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (CVA) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Chest pain - Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dizziness (General disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fluid volume overload( i.e. diuresis, electrolyte imbalance) (Ablation Procedure) (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 5 (5) | 4 (4) | 2 (3) | 0 (0)
Genitourinary (Renal and urinary disorders) | 8 (9) | 1 (1) | 0 (0) | 0 (0)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 3 (3) | 2 (2) | 3 (4) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart failure symptoms - Unspecified (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Hematoma (Ablation Procedure) (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hiccups (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
IV infiltrate (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple heart failure symptoms (Cardiac disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Multiple symptoms (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 9 (9) | 3 (3) | 2 (2) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Other SVT (AVRT, AVNRT, EAT etc. (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericardial Effusion (Ablation Procedure) (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Ablation Procedure) (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Premature atrial contractions (PAC) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Psychological (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 7 (8) | 1 (1) | 0 (0)
Pulmonary Vein Stenosis - Significant (>70%) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary edema - Heart failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (PE) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectus sheath hematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Renal insufficiency - Heart failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sanguineous drainage (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blazer Open-Irrigated Ablation Catheter Randomized (N=159) | FDA Approved Open-Irrigated Ablation Catheter Randomized (N=167) | Blazer Open-Irrigated Ablation Catheter Roll-In (N=51) | FDA Approved Open-Irrigated Ablation Catheter Roll-In (N=1)
1st degree AV block (Cardiac disorders) | 7 (7) | 5 (5) | 0 (0) | 0 (0)
2nd degree AV block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AV Fistula (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal laboratory values (General disorders) | 6 (6) | 1 (1) | 2 (2) | 0 (0)
Adverse medication reaction (General disorders) | 9 (11) | 8 (8) | 3 (3) | 0 (0)
Allergic reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Ablation Procedure) (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anesthesia/Sedation related complication (Ablation Procedure) (General disorders) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Angina (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic root atheromatosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Ablation Procedure) (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arterial/Venous Thromboembolic Events (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (AF) (Cardiac disorders) | 22 (22) | 32 (33) | 12 (12) | 0 (0)
Atrial flutter (type 1 Isthmus Dependent) (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2) | 0 (0)
Atrial tachycardia (Cardiac disorders) | 11 (11) | 6 (6) | 0 (0) | 0 (0)
Atypical Atrial Flutter (Cardiac disorders) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Back discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bradycardia with pauses (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breathing difficulties (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brugada syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 12 (13) | 6 (9) | 3 (3) | 0 (0)
Chest pain - Ischemic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cirrhosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cyst on ascending aorta (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Difficulty sleeping (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (General disorders) | 2 (2) | 7 (7) | 2 (2) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 1 (1) | 0 (0)
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (Ablation Procedure) (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exacerbation of existing condition (Ablation Procedure) (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fluid retention (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 9 (10) | 9 (12) | 3 (3) | 0 (0)
Gastroparesis (Ablation Procedure) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genitourinary (Renal and urinary disorders) | 10 (10) | 10 (10) | 4 (4) | 0 (0)
Groin bleed (Ablation Procedure) (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 13 (13) | 12 (14) | 3 (3) | 0 (0)
Heart failure symptoms - Unspecified (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hematological (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Ablation Procedure) (Vascular disorders) | 7 (7) | 4 (4) | 4 (4) | 0 (0)
Hemorrhage (Ablation Procedure) (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 5 (6) | 3 (3) | 1 (1) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Ablation Procedure) (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Integumentary (General disorders) | 5 (5) | 3 (3) | 1 (1) | 0 (0)
Intracardiac thrombus with no thromboembolic event (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Intraventricular conduction delay (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Junctional ectopic rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Long QT (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Multiple heart failure symptoms (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 7 (7) | 8 (8) | 2 (2) | 0 (0)
Neurological (Nervous system disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0)
Non-toxic LLE cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nonsustained ventricular tachycardia (NSVT) (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Other SVT (AVRT, AVNRT, EAT etc. (Cardiac disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Pain neuromuscular/non cardiovascular (Ablation Procedure) (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 4 (4) | 6 (7) | 2 (2) | 0 (0)
Pericardial Effusion (Ablation Procedure) (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion - Unrelated to procedure (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Peripheral edema (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Peripheral edema - Heart failure (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Physical trauma (General disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Pleuritis (Ablation Procedure) (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Premature atrial contractions (PAC) (Cardiac disorders) | 5 (5) | 2 (2) | 1 (1) | 0 (0)
Premature ventricular contractions (PVC) (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Pseudoaneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychological (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 9 (9) | 1 (2) | 0 (0)
Pulmonary Vein Stenosis - Mild or Moderate (<70%) (Cardiac disorders) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
Pulmonary Vein Stenosis - Significant (>70%) (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Renal (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Right bundle branch block (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 5 (5) | 6 (6) | 2 (2) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 8 (8) | 4 (4) | 0 (0) | 0 (0)
Sore throat (General disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Swollen groin (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Syncope (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Ablation Procedure) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombus (No embolism) (Ablation Procedure) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Typical atrial flutter (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vagal denervation symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (VT) (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual Blurring/Disturbances (Ablation Procedure) (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other